CLINICAL TRIAL: NCT04543188
Title: A TWO-PART, PHASE 1A/B, OPEN-LABEL, MULTICENTER TRIAL EVALUATING PHARMACOKINETICS, SAFETY AND EFFICACY OF PF 07284890 (ARRY 461) IN PARTICIPANTS WITH BRAF V600 MUTANT SOLID TUMORS WITH AND WITHOUT BRAIN INVOLVEMENT
Brief Title: A FIH Study of PF-07284890 in Participants With BRAF V600 Mutant Solid Tumors With and Without Brain Involvement
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Pfizer has made an internal business decision to not continue further development of PF-07284890. This decision was not due to major safety concerns or requests from any regulatory authorities.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4471001; 2022-003184-23 (EudraCT Number)
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Malignant Melanoma; Carcinoma, Non-Small-Cell Lung; Brain Neoplasms, Primary; Brain Neoplasms; Malignant Neoplasms
Keywords: Proto-Oncogene Proteins B-raf; Brain Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung; Brain Diseases; Central Nervous System Neoplasms; Enzyme Inhibitors
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Neoplasms; Brain Diseases; Central Nervous System Neoplasms | interventions — PF-07284890; binimetinib; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- PF-07284890 (Part A monotherapy) (Experimental): Monotherapy dose escalation of PF-07284890
  Interventions: Drug: PF-07284890
- PF-07284890+binimetinib (Part A combo-therapy) (Experimental): Combination dose escalation of PF-07284890 + binimetinib
  Interventions: Drug: PF-07284890; Drug: Binimetinib
- Expansion Phase (Part B, Cohort 1) (Experimental): PF-07284890 (at recommended dose from Part A) plus binimetinib in participants with BRAF V600 melanoma, with asymptomatic brain involvement, and no prior BRAF or MEK inhibitor utilization
  Interventions: Drug: PF-07284890; Drug: Binimetinib
- Expansion Phase (Part B, Cohort 2) (Experimental): PF-07284890 (at recommended dose from Part A) plus binimetinib in participants with BRAF V600 melanoma, with symptomatic brain involvement, and no prior BRAF or MEK inhibitor utilization
  Interventions: Drug: PF-07284890; Drug: Binimetinib
- Expansion Phase (Part B, Cohort 3) (Experimental): PF-07284890 (at recommended dose from Part A) plus binimetinib in participants with BRAF V600 melanoma, with asymptomatic brain involvement, and prior BRAF inhibitor utilization
  Interventions: Drug: PF-07284890; Drug: Binimetinib
- Expansion Phase (Part B, Cohort 4) (Experimental): PF-07284890 (at recommended dose from Part A) plus binimetinib in participants with BRAF V600 melanoma, with symptomatic brain involvement, and prior BRAF inhibitor utilization
  Interventions: Drug: PF-07284890; Drug: Binimetinib
- Expansion Phase (Part B Cohort 5) (Experimental): PF-07284890 (at recommended dose from Part A) plus binimetinib in participants with BRAF V600 solid tumor; history of or current leptomeningeal metastases; without disease in the brain; with disease in the brain that does not meet Cohorts 1-4; asymptomatic or symptomatic in the brain; primary brain tumors
  Interventions: Drug: PF-07284890; Drug: Binimetinib
- Expansion Phase Drug-Drug Interaction Substudy (Part B Optional Cohort 6) (Experimental): PF-07284890 (at recommended dose from Part A) plus binimetinib plus midazolam in participants with BRAF V600 solid tumor
  Interventions: Drug: PF-07284890; Drug: Binimetinib; Drug: Midazolam
- Expansion Phase (Part B Optional Cohort 7) (Experimental): PF-07284890 (at the recommended dose for expansion when administered with food) plus binimetinib in participants with BRAF V600 solid tumor
  Interventions: Drug: PF-07284890; Drug: Binimetinib

INTERVENTIONS:
Drug: PF-07284890 — PF-07284890 will be administered orally, daily for 21 consecutive days (21-day cycle)
  Other Names: ARRY-461
Drug: Binimetinib — Binimetinib will be administered together with PF-07284890 orally, 45mg twice daily
  Other Names: Mektovi
  Arms: Expansion Phase (Part B Cohort 5); Expansion Phase (Part B Optional Cohort 7); Expansion Phase (Part B, Cohort 1); Expansion Phase (Part B, Cohort 2); Expansion Phase (Part B, Cohort 3); Expansion Phase (Part B, Cohort 4); Expansion Phase Drug-Drug Interaction Substudy (Part B Optional Cohort 6); PF-07284890+binimetinib (Part A combo-therapy)
Drug: Midazolam — Midazolam will be administered 7 days before start of study drug, on Cycle 1 Day 1, and on Cycle 1 Day 15
  Arms: Expansion Phase Drug-Drug Interaction Substudy (Part B Optional Cohort 6)

SUMMARY:
First-in-human study to assess safety, tolerability, PK, and preliminary activity of PF-07284890 as a single agent and in combination with binimetinib in participants with BRAF V600-mutated advanced solid tumor malignancies with and without brain involvement.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16 years at the time of consent
* Histologically confirmed diagnosis of advanced/metastatic solid tumor including primary brain tumor
* Documented evidence of a BRAF V600 mutation in tumor tissue or blood
* Confirmation of availability of adequate tumor tissue for submission to the sponsor/central laboratory
* Presence or absence of brain involvement unless specified below
* Dose Expansion (Part B)

  * Cohort 1, 2, 3, 4: melanoma with at least 1 parenchymal brain lesion
  * Cohort 1,3: asymptomatic in the brain for at least 14 days prior to start of study treatment
  * Cohort 2,4: symptomatic in the brain within 14 days prior to the start of study treatment
  * Cohort 5: any solid tumor that does not meet requirements for Cohorts 1-4, history of or current leptomeningeal metastases.
  * Optional Cohort 6 (DDI Sub-study) and 7 (Food-Effect): if brain involvement present, must be asymptomatic
* Disease progression despite prior treatment and no acceptable alternative treatment options available unless specified below
* Dose Expansion (Part B)

  * Cohort 1, 2: No prior BRAF inhibitor in the metastatic setting or in the adjuvant setting within 6 months of study treatment
  * Cohort 3, 4: Required prior BRAF inhibitor in the metastatic setting or in the adjuvant setting within 6 months of treatment
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1

Exclusion Criteria:

* Brain metastasis/primary brain tumor requiring immediate local intervention
* History of or current leptomeningeal metastases
* Any other active malignancy within 2 years prior to enrollment
* Radiation therapy to visceral metastases within 14 days prior to study treatment. WBRT within 28 days prior to study treatment.
* Systemic anti-cancer therapy or small-molecular therapeutic(s) within 2 weeks prior to start of study treatment; Antibody based agents within 4 weeks prior to start of study treatment.
* History or current evidence of RVO or current risk factors for RVO; History of retinal degenerative disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (39):
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Richard M Schulze Family Foundation Outpatient Center at McKinley Campus, Tampa, Florida
  - Northwestern Medical Group, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Johns Hopkins University / Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ophthalmic Consultants of Boston Inc (OCB), Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Imaging: Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Imaging: Brigham and Women's Radiology, Coolidge Corner Imaging, Brookline, Massachusetts
  - Imaging: Brigham and Women's Ambulatory Care, Chestnut Hill, Massachusetts
  - Imaging: Brigham and Women's Mass General Healthcare Center, Foxborough, Massachusetts
  - Dana-Farber Cancer Institute - Chestnut Hill, Newton, Massachusetts
  - Siteman Cancer Center - St Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Siteman Cancer Center - North County, Florissant, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - MSK Monmouth., Middletown, New Jersey
  - MSK Commack, Commack, New York
  - MSKCC-Westchester (500 Westchester Ave.), Harrison, New York
  - Memorial Sloan Kettering Cancer Center - David H. Koch Center for Cancer Care (74th Street)., New York, New York
  - Rockefeller Outpatient Pavilion (53rd Street), New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Eye Center, Durham, North Carolina
  - Duke University Medical Center, Investigational Chemotherapy Services, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Tennessee Oncology PLLC, Franklin, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Israel (5):
  - Rambam Health Care Campus, Haifa, ?eif?
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Sourasky Medical Center, Tel Aviv, TELL ABĪB

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Ren L, Moreno D, Baer BR, Barbour P, Bettendorf T, Bouhana K, Brown K, Brown SA, Fell JB, Hartley DP, Hicken EJ, Laird ER, Lee P, McCown J, Otten JN, Prigaro B, Wallace R, Kahn D. Identification of the Clinical Candidate PF-07284890 (ARRY-461), a Highly Potent and Brain Penetrant BRAF Inhibitor for the Treatment of Cancer. J Med Chem. 2024 Aug 8;67(15):13019-13032. doi: 10.1021/acs.jmedchem.4c00998. Epub 2024 Jul 30. PMID 39077892
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4471001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of 2 phases: Phase 1a (dose escalation, divided into monotherapy [PF-07284890 alone] and combination therapy [PF-07284890 plus binimetinib]) and Phase 1b (dose expansion).
Pre-assignment Details: A total of 65 participants were enrolled in the study: Phase 1a: 48 participants (monotherapy [25 participants] and combination therapy [23 participants]) and Phase 1b: 17 participants). No participants were enrolled in Cohort 2 and 6 of Phase 1b.
Groups:
- Phase 1a: PF-07284890 50 mg QD: Participants received PF-07284890 50 milligrams (mg) oral dose once daily (QD) in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 100 mg QD: Participants received PF-07284890 100 mg oral dose QD in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 200 mg QD: Participants received PF-07284890 200 mg oral dose QD in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 200 mg BID: Participants received PF-07284890 200 mg oral dose twice daily (BID) in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 300 mg BID: Participants received PF-07284890 300 mg oral dose BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 450 mg BID: Participants received PF-07284890 450 mg oral dose BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID: Participants received PF-07284890 100 mg oral dose QD in combination with binimetinib 45 mg oral dose BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID: Participants received PF-07284890 100 mg oral dose BID in combination with binimetinib 45 mg oral dose BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID: Participants received PF-07284890 150 mg oral dose BID in combination with binimetinib 45 mg oral dose BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID: Participants received PF-07284890 225 mg oral dose BID in combination with binimetinib 45 mg oral dose BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID: Participants received PF-07284890 300 mg oral dose BID in combination with binimetinib 45 mg oral dose BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1b: Cohort 1: Cohort 1 included melanoma participants with asymptomatic brain metastases and no prior B-type Raf proto-oncogene (BRAF) inhibitor therapy. Participants received PF-07284890 300 mg oral dose QD in combination with binimetinib 45 mg BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1b: Cohort 3: Cohort 3 included melanoma participants with asymptomatic brain metastases and with prior BRAF inhibitor therapy. Participants received PF-07284890 300 mg oral dose QD in combination with binimetinib 45 mg BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1b: Cohort 4: Cohort 4 included melanoma participants with symptomatic brain metastases and with prior BRAF inhibitor therapy. Participants received PF-07284890 300 mg oral dose QD in combination with binimetinib 45 mg BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1b: Cohort 5: Cohort 5 included participants with a mixture of tumor types, any brain disease and with or without prior BRAF inhibitor therapy. Participants received PF-07284890 300 mg oral dose QD in combination with binimetinib 45 mg BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
Period: Phase 1a
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Started | 2 | 4 | 3 | 3 | 10 | 3 | 4 | 4 | 2 | 5 | 8 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 4 | 3 | 3 | 10 | 3 | 4 | 4 | 2 | 5 | 8 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other (Death) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 2 | 2 | 3 | 1 | 4 | 2 | 3 | 4 | 1 | 0 | 4 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Global Deterioration Of Health Status | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Phase 1b
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 11
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Other (Death) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 5
Not completed — Study Terminated By Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set included all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5 | Total
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 10 | 3 | 4 | 4 | 2 | 5 | 8 | 1 | 4 | 1 | 11 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (0.71) | 56.3 (12.61) | 65.3 (12.34) | 62.7 (11.85) | 55.9 (15.95) | 50.0 (7.94) | 59.8 (3.20) | 57.5 (23.35) | 40.5 (27.58) | 42.0 (18.71) | 45.0 (13.89) | 57.0 (NA) — Standard deviation (SD) could not be calculated as only 1 participant was available for analysis. | 63.8 (12.15) | 31.0 (NA) — SD could not be calculated as only 1 participant was available for analysis. | 50.8 (12.96) | 53.4 (15.12)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 0 | 3 | 3 | 1 | 3 | 0 | 3 | 1 | 1 | 4 | 4 | 0 | 1 | 0 | 6 | 30
  Female | 2 | 1 | 0 | 2 | 7 | 3 | 1 | 3 | 1 | 1 | 4 | 0 | 3 | 0 | 5 | 33
  Not disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 4 | 3 | 3 | 9 | 3 | 3 | 4 | 2 | 3 | 7 | 0 | 4 | 0 | 9 | 56
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Not reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 5
  Not disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/ Latino(a) or of Spanish Origin | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 5
  Not Hispanic/Latino(a)/of Spanish Origin | 2 | 3 | 3 | 3 | 8 | 3 | 4 | 4 | 2 | 4 | 6 | 0 | 4 | 0 | 11 | 57
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs): Phase 1a
Description: DLT was defined as any adverse event (AE) or abnormal laboratory value which were related to study treatment and assessed as unrelated to disease (disease progression), occurring during the first 21 days of treatment that met at least 1 of the study specified criteria. DLTs were graded according to the National Cancer Institute- Common Terminology Criteria for Adverse Events (NCI-CTCAE), version (v) 5.0.
Time Frame: Cycle 1 (21 Days)
Population: The per protocol analysis set included all enrolled participants who had at least one dose of study treatment and either experienced DLT or did not have major treatment deviations during the DLT observation period.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID: Participants received PF- 07284890 150 mg oral dose BID in combination with binimetinib 45 mg oral dose BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 3 | 3 | 2 | 6 | 1 | 4 | 3 | 2 | 3 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, Serious Treatment Related TEAEs, Grade 3 or 4 TEAEs and Grade 5 TEAEs by NCI CTCAE v5.0: Phase 1a
Description: An adverse event (AE) was any untoward medical occurrence in participant/ clinical study participant temporally associated with use of study intervention, whether/ not considered related to study intervention. TEAEs were defined as any AE that occurs during on-treatment period. The on-treatment period was defined as period that starts with first dose of study treatment and ends at last dose of study treatment +30 days, or start of new anti-cancer therapy [- 1 day], whichever occurred first. Serious TEAEs were any untoward medical occurrence at any dose that: suspected to cause death; life-threatening; required hospitalization; persistent/significant disability/incapacity and might caused congenital anomaly/birth defect. Serious treatment related TEAEs were related to study treatment and relatedness was judged by investigator. TEAEs were graded according to NCI-CTCAE v 5.0 (grade 3= severe, grade 4= life-threatening and grade 5= death related to AE). AEs included SAEs and all non-SAE.
Time Frame: From first dose of study treatment (Day 1) up to 30 days post last dose of study treatment or start of new anti-cancer therapy (-1 Day) whichever occurred first (maximum treatment exposure: 542 days; maximum follow-up: 572 days)
Population: The safety analysis set included all enrolled participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 10 | 3 | 4 | 4 | 2 | 5 | 8
Participants
  Participants with TEAEs | 2 | 4 | 3 | 3 | 10 | 3 | 4 | 4 | 2 | 5 | 8
  Participants with Serious TEAEs | 0 | 1 | 0 | 3 | 4 | 2 | 1 | 1 | 1 | 2 | 3
  Participants with serious treatment related TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Participants with Grade 3 or 4 TEAEs | 1 | 1 | 0 | 2 | 5 | 0 | 3 | 4 | 1 | 1 | 3
  Participants with Grade 5 TEAEs | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 2

3. Primary Outcome: Number of Participants With Hematology Laboratory Abnormalities of Any CTCAE Grade: Phase 1a
Description: The following hematology laboratory parameters were assessed: activated partial thromboplastin time prolonged, anemia, hemoglobin increased, international normalized ratio (INR) increased, leukocytosis, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased and white blood cell decreased. Laboratory abnormality events were graded according to NCI CTCAE v5.0; grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening consequences and grade 5=death. In this outcome measure, those number of participants are reported who had hematology laboratory abnormality in any parameter of any CTCAE Grades.
Time Frame: From first dose of study treatment (Day 1) up to 30 days post last dose of study treatment (maximum treatment exposure: 542 days; maximum follow-up: 572 days)
Population: The safety analysis set included all enrolled participants who received at least one dose of study intervention. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 10 | 2 | 4 | 4 | 2 | 5 | 8
Participants | 2 | 4 | 3 | 3 | 10 | 2 | 4 | 4 | 2 | 5 | 8

4. Primary Outcome: Number of Participants With Chemistry Laboratory Abnormalities of Any CTCAE Grade: Phase 1a
Description: The following chemistry laboratory parameters were assessed: alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, creatine phosphokinase (CPK) increased, creatinine increased, hypercalcemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia and hyponatremia. Laboratory abnormality events were graded according to NCI CTCAE v5.0; grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening consequences and grade 5=death. In this outcome measure, those number of participants are reported who had chemistry laboratory abnormality in any parameter of any CTCAE Grades.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 10 | 2 | 4 | 4 | 2 | 5 | 8
Participants | 2 | 4 | 3 | 3 | 10 | 2 | 4 | 4 | 2 | 5 | 8

5. Primary Outcome: Number of Participants With Dose Interruptions Due to TEAEs: Phase 1a
Description: Dose interruption was defined as a planned dosing day with 0 mg total dose administered. Dose interruptions were applicable to unexpected dose interruptions. In this outcome measure, dose interruptions for any drug were considered.
Time Frame: During study treatment (from first dose of study treatment [Day 1] up to last dose of study treatment [maximum treatment exposure: 542 days])
Population: The safety analysis set included all enrolled participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 10 | 3 | 4 | 4 | 2 | 5 | 8
Participants | 0 | 1 | 0 | 3 | 5 | 1 | 2 | 3 | 1 | 2 | 5

6. Primary Outcome: Number of Participants With Dose Reduction Due to TEAEs: Phase 1a
Description: A dose reduction was defined as the day when the actual dose was less than the planned dose at enrollment and the actual dose was greater than 0 mg (ie, missed doses were not counted as a reduction). In this outcome measure, dose reductions for any drug were considered.
Time Frame: as for outcome 5
Population: The safety analysis set included all enrolled participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 10 | 3 | 4 | 4 | 2 | 5 | 8
Participants | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 2

7. Primary Outcome: Number of Participants With Dose Discontinuations Due to TEAEs: Phase 1a
Description: In this outcome measure, dose discontinuations for any drug due to TEAEs were considered.
Time Frame: as for outcome 5
Population: The safety analysis set included all enrolled participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 10 | 3 | 4 | 4 | 2 | 5 | 8
Participants | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 1

8. Primary Outcome: Extracranial Response Rate by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1: Phase 1b
Description: Extracranial response rate was defined as the percentage of participants with a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) in extracranial lesions by Investigator assessment per RECIST v1.1. CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (non-target) must have reduction in short axis to less than (<) 10 millimeter (mm). PR: at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of first dose until CR or PR (maximum treatment exposure: 400 days)
Population: Extracranial response evaluable set included all participants enrolled and received at least one dose of study treatment and had measurable tumor at baseline and at least one post baseline extracranial assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 1 | 1 | 8
Percentage of participants | 100.0 [2.5 to 100.0] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 12.5 [0.3 to 52.7]

9. Primary Outcome: Intracranial Response Rate by mRECISTv1.1: Phase 1b
Description: Intracranial response rate as assessed using modified RECIST (mRECIST) v 1.1., was defined as the percentage of participants with brain or central nervous system (CNS) involvement who achieved a CR or PR. CR: disappearance of all target and non-target lesions. For target lesions: Any pathological lymph nodes must be <10 mm in the short axis. For non-target lesions: All lymph nodes identified as a site of disease at baseline must be non-pathological (eg, <10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of first dose until CR or PR (maximum treatment exposure: 400 days)
Population: Intracranial response evaluable set included all participants enrolled and received at least one dose of study treatment and had measurable brain tumor at baseline and at least one post baseline intracranial assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 2 | 1 | 3
Percentage of participants | 0 [0.0 to 97.5] | 0 [0.0 to 84.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]

10. Primary Outcome: Overall Response Rate (ORR): Phase 1b
Description: ORR: percentage of participants with BOR of confirmed CR/PR by investigator assessment in intracranial metastasis (mRECISTv1.1) and extracranial lesions (RECISTv1.1). RECIST v1.1- CR: disappearance of all target and non-target lesions. Any pathological lymph node (non-target) must have reduction in short axis to <10mm. PR: at least 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters. mRECIST- CR: disappearance of all target and non-target lesion. For target lesion: Any pathological lymph nodes must be <10 mm in short axis. For non-target lesion: All lymph nodes identified as site of disease at baseline must be non-pathological (eg, <10 mm short axis). PR: at least 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters.
Time Frame: From date of first dose until CR or PR (maximum treatment exposure: 400 days)
Population: The response evaluable population included all participants who received at least one dose of study treatment and had measurable disease at baseline and at least one post baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 1 | 1 | 9
Percentage of participants | 100 [2.5 to 100.0] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 11.1 [0.3 to 48.2]

11. Primary Outcome: Response Rate Using Response Assessment in Neuro-Oncology (RANO) for Primary Brain Tumors: Phase 1b
Description: RANO response rate was defined as the percentage of glioblastoma participants who achieved a CR or PR per RANO. CR was defined as complete disappearance of all enhancing measurable and non-measurable disease sustained for more than or equal to (>=) 4 weeks; no new lesions; stable or improved non-enhancing (T2/ [fluid attenuated inversion recovery] FLAIR) lesions; off steroids and neurological condition stable or improved. PR was defined as >=50% decrease compared to baseline in the sum of the perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks; no progression of non-measurable disease; no new lesions; stable or improved non enhancing (T2/FLAIR) lesions on the same or lower dose of corticosteroids compared with baseline scan; the corticosteroid dose at the time of the scan evaluation should be no greater than the dose at the time of the baseline scan and neurological condition stable or improved.
Time Frame: From date of first dose until CR or PR (maximum treatment exposure: 400 days)
Population: The response evaluable population analyzed. The outcome measure was to be evaluated only in glioblastoma participants; apart from Cohort 5 all other cohorts did not have any glioblastoma participants. Hence, "Overall Number of Participants Analyzed" for these cohorts is "0" and for Cohort 5 it signifies participants evaluable for this outcome.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 0 | 0 | 0 | 2
Percentage of participants |  |  |  | 50.0 [1.3 to 98.7]

12. Secondary Outcome: Maximum Observed Concentration (Cmax) of PF-07284890 and Binimetinib for Single Dose: Phase 1a
Time Frame: Pre-dose,1, 2, 4, 6, 8 and 24 hours post-dose on Cycle 1 Day 1 (C1D1); 24 hours was only for arms where study drug was administered as QD.
Population: The pharmacokinetic (PK) parameter analysis population included all enrolled participants treated who did not have protocol deviations influencing PK parameter assessment and have sufficient information to estimate at least 1 of the PK parameters of interest.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 10 | 3 | 4 | 4 | 2 | 5 | 6
Nanogram per milliliter (ng/mL)
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 549 and 1040 ng/mL. | 1692 (541.62) | 1603 (308.92) | 1983 (789.96) | 2466 (1008.9) | 1771 (1360.5) | 1893 (968.86) | 2009 (922.45) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 2350 and 3220 ng/mL. | 3286 (1539.4) | 2339 (1220.8)
  Binimetinib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 1 | 5 | 5
  Binimetinib |  |  |  |  |  |  | 432.3 (153.53) | 457.5 (174.37) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 329 ng/mL. | 396.2 (208.55) | 287.0 (127.42)

13. Secondary Outcome: Time for Cmax (Tmax) of PF-07284890 and Binimetinib for Single Dose: Phase 1a
Time Frame: Pre-dose,1, 2, 4, 6, 8 and 24 hours post-dose on C1D1; 24 hours was only for arms where study drug was administered as QD.
Population: The PK parameter analysis population included all enrolled participants treated who did not have protocol deviations influencing PK parameter assessment, and have sufficient information to estimate at least 1 of the PK parameters of interest. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and contributed to data; 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 10 | 3 | 4 | 4 | 2 | 5 | 6
Hours
  PF-07284890 | NA [NA to NA] — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence median and full range not reported. Individual values were 1.00 and 2.18 hours. | 4.94 [2.07 to 5.93] | 5.93 [2.32 to 6.18] | 5.87 [4.08 to 5.97] | 3.95 [1.00 to 6.00] | 2.00 [1.02 to 6.02] | 3.44 [0.817 to 22.8] | 4.00 [2.45 to 7.83] | NA [NA to NA] — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence median and full range not reported. Individual values were 1.85 and 5.85 hours. | 3.92 [2.00 to 7.70] | 3.12 [0.967 to 7.73]
  Binimetinib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 1 | 5 | 5
  Binimetinib |  |  |  |  |  |  | 1.01 [0.817 to 2.12] | 1.66 [1.00 to 2.07] | NA [NA to NA] — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence median and full range not reported. Individual value was 2.03 hours. | 1.00 [1.00 to 2.08] | 1.00 [0.967 to 2.07]

14. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to the Last Time Point of Quantifiable Concentration (AUClast) of PF-07284890 and Binimetinib for Single Dose: Phase 1a
Description: AUClast was determined using the linear/log trapezoidal method.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 10 | 3 | 4 | 4 | 2 | 5 | 6
Nanogram*hour per milliliter (ng*hr/mL)
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 8330 and 9100 ng*hr/mL. | 14960 (6415.5) | 16400 (3404.4) | 8883 (6085.0) | 13250 (6943.8) | 8883 (8251.1) | 21920 (15893) | 9858 (5391.9) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 10800 and 17900 ng*hr/mL. | 17090 (7615.8) | 11270 (5458.1)
  Binimetinib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 1 | 5 | 5
  Binimetinib |  |  |  |  |  |  | 1710 (1362.5) | 1639 (673.91) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 1490 ng*hr/mL. | 1289 (358.45) | 979.4 (227.90)

15. Secondary Outcome: Terminal Elimination Half Life (t½) of PF-07284890 and Binimetinib for Single Dose: Phase 1a
Description: T1/2 was calculated as loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: as for outcome 13
Population: The PK parameter analysis population used. Here "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure and contributed to data; 'Number Analyzed' =number of participants evaluable for specified rows. T1/2 could not be calculated for all participants due to challenges with determining T1/2 using an 8-hour profile particularly for C1D1 (where the pre-dose sample cannot be used), so the data could not be included and thus reported as 0 as applicable.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 1 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 3 | 4
Hours
  PF-07284890: number analyzed (Participants) | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 6.39 hours. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 5.89 and 7.25 hours. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 5.83 hours. |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 2.45 hours. |  |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 2.60 hours. |  |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 2.42 hours.
  Binimetinib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 3 | 4
  Binimetinib |  |  |  |  |  |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 1.70 and 2.44 hours. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 2.48 hours. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 1.77 hours. | 2.153 (0.62389) | 2.443 (0.91318)

16. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero Extrapolated to Infinity (AUCinf) of PF-07284890 and Binimetinib for Single Dose: Phase 1a
Description: AUCinf was calculated as AUClast + (Clast/kel), where Clast is the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis. Those outcome measures are either due to either patient(s) has insufficient sample(s) (e.g., sampling only through Tmax or 1 sample after) for analyses or t1/2 could not be determined
Time Frame: as for outcome 13
Population: PK parameter analysis population used. "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure and contributed to data; 'Number Analyzed' =number of participants evaluable for specified rows. AUCinf could not be calculated either due to either participants had insufficient sample(s) (e.g., sampling only through Tmax or 1 sample after) for analyses or t1/2 could not be determined, which affects the ability to calculate AUCinf and thus reported 0 as applicable.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 1 | 2 | 1 | 0 | 2 | 1 | 3 | 4 | 1 | 5 | 5
ng*hr/mL
  PF-07284890: number analyzed (Participants) | 1 | 2 | 1 | 0 | 2 | 1 | 1 | 1 | 1 | 1 | 3
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 8990 ng*hr/mL. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 10200 and 14900 ng*hr/mL. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 68500 ng*hr/mL. |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 8030 and 12600 ng*hr/mL. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 17200 ng*hr/mL. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 11200 ng*hr/mL. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 9610 ng*hr/mL. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 14000 ng*hr/mL. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 29000 ng*hr/mL. | 15390 (9558.0)
  Binimetinib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 1 | 5 | 5
  Binimetinib |  |  |  |  |  |  | 3128 (3244.1) | 1958 (871.79) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 1630 ng*hr/mL. | 1643 (631.36) | 1437 (628.11)

17. Secondary Outcome: Apparent Oral Clearance (CL/F) of PF-07284890 and Binimetinib for Single Dose: Phase 1a
Description: CL/F was calculated as Dose/AUCinf.
Time Frame: as for outcome 13
Population: PK parameter analysis population used. "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure and contributed to data; 'Number Analyzed' =number of participants evaluable for specified rows. CL/F could not be calculated either due to either participants had insufficient sample(s) (e.g., sampling only through Tmax or 1 sample after) for analyses or t1/2 could not be determined, which affects the ability to calculate CL/F and thus reported 0 as applicable.
Measure: Mean (Standard Deviation); unit: Liter per hour (L/hr)
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 1 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 3 | 4
Liter per hour (L/hr)
  PF-07284890: number analyzed (Participants) | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 5.56 L/hr. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 6.71 and 9.77 L/hr. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 11.6 L/hr. |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 23.9 L/hr. |  |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 10.4 L/hr. |  |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 28.5 L/hr.
  Binimetinib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 3 | 4
  Binimetinib |  |  |  |  |  |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 25.5 and 57.5 L/hr. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 26.1 L/hr. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 27.6 L/hr. | 33.97 (13.627) | 40.48 (12.458)

18. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-07284890 and Binimetinib for Single Dose: Phase 1a
Description: Vz/F was calculated as Dose/(AUCinf * kel) where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: as for outcome 13
Population: PK parameter analysis population used. "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure and contributed to data; 'Number Analyzed' =number of participants evaluable for specified rows. Vz/F could not be calculated either due to either participants had insufficient sample(s) (e.g., sampling only through Tmax or 1 sample after) for analyses or t1/2 could not be determined, which affects the ability to calculate Vz/F and thus reported 0 as applicable.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 1 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 3 | 4
Liter
  PF-07284890: number analyzed (Participants) | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 51.3 L. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 57.1 and 102 L. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 97.8 L. |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 84.3 L. |  |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 39.0 L. |  |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 99.7 L.
  Binimetinib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 3 | 4
  Binimetinib |  |  |  |  |  |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 89.7 and 141 L. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 93.4 L. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 70.5 L. | 97.50 (7.1757) | 139.3 (52.043)

19. Secondary Outcome: Cmax of PF-07284890 and Binimetinib for Multiple Dose: Phase 1a
Time Frame: Pre-dose,1, 2, 4, 6 and 8 hours post dose on C1D15
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 3 | 3 | 2 | 7 | 1 | 3 | 4 | 2 | 4 | 6
ng/mL
  PF-0728489 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 943 and 1940 ng/mL. | 1102 (178.49) | 1830 (291.03) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 2610 and 4870 ng/mL. | 3489 (1647.2) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 1070 ng/mL. | 1991 (1325.5) | 2270 (844.63) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 1970 and 3800 ng/mL. | 3870 (655.34) | 3613 (739.91)
  Binimetinib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 2 | 4 | 6
  Binimetinib |  |  |  |  |  |  | 518.3 (243.47) | 633.8 (370.06) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 534 and 732 ng/mL. | 674.0 (276.30) | 457.3 (180.50)

20. Secondary Outcome: Tmax of PF-07284890 and Binimetinib for Multiple Dose: Phase 1a
Time Frame: Pre-dose,1, 2, 4, 6 and 8 hours post dose on C1D15
Population: as for outcome 13
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 3 | 3 | 2 | 7 | 1 | 3 | 4 | 2 | 4 | 6
Hours
  PF-07284890 | NA [NA to NA] — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence median and full range not reported. Individual values were 1.00 and 2.02 hours. | 4.03 [2.00 to 4.13] | 2.15 [2.08 to 4.03] | NA [NA to NA] — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence median and full range not reported. Individual values were 2.20 and 4.13 hours. | 3.90 [1.05 to 5.75] | NA [NA to NA] — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence median and full range not reported. Individual values was 1.07 hours. | 3.95 [2.05 to 7.80] | 2.08 [2.03 to 4.00] | NA [NA to NA] — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence median and full range not reported. Individual values were 2.22 and 3.92 hours. | 2.01 [2.00 to 4.00] | 2.03 [0.983 to 3.92]
  Binimetinib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 2 | 4 | 6
  Binimetinib |  |  |  |  |  |  | 1.93 [1.00 to 7.80] | 0.977 [0.000 to 2.40] | NA [NA to NA] — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence median and full range not reported. Individual values were 0.950 and 1.85 hours. | 1.01 [1.00 to 1.92] | 1.04 [0.967 to 2.25]

21. Secondary Outcome: Area Under the Plasma Concentration Time Curve Over the Dosing Interval (AUCtau) of PF-07284890 and Binimetinib for Multiple Dose: Phase 1a
Time Frame: Pre-dose,1, 2, 4, 6 and 8 hours post dose on C1D15
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 3 | 3 | 2 | 7 | 1 | 3 | 4 | 2 | 4 | 6
ng*hr/mL
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 10600 and 12300 ng*hr/mL. | 10260 (813.65) | 16530 (1616.6) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 15200 and 47600 ng*hr/mL. | 30030 (16644) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 6630 ng*hr/mL. | 15370 (5218.1) | 17450 (7857.3) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 14300 and 32800 ng*hr/mL. | 28550 (5569.3) | 29400 (9041.5)
  Binimetinib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 2 | 4 | 6
  Binimetinib |  |  |  |  |  |  | 2740 (1196.2) | 3150 (1749.5) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 1880 and 4610 ng*hr/mL. | 2458 (341.89) | 2420 (1306.5)

22. Secondary Outcome: Lowest Concentration Observed During the Dosing Interval (Cmin) of PF-07284890 and Binimetinib for Multiple Dose: Phase 1a
Time Frame: Pre-dose,1, 2, 4, 6 and 8 hours post dose on C1D15
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 3 | 3 | 2 | 7 | 1 | 3 | 4 | 2 | 4 | 6
ng/mL
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 137 and 195 ng/mL. | 130.2 (67.258) | 198.0 (155.75) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 267 and 3270 ng/mL. | 1773 (1344.9) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 351 ng/mL. | 181.7 (99.887) | 822.3 (441.12) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 435 and 1290 ng/mL. | 1223 (602.84) | 1625 (612.23)
  Binimetinib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 2 | 3 | 6
  Binimetinib |  |  |  |  |  |  | 73.57 (28.576) | 127.1 (66.662) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 82.3 and 269 ng/mL. | 67.13 (26.085) | 94.72 (32.053)

23. Secondary Outcome: CL/F of PF-07284890 and Binimetinib for Multiple Dose: Phase 1a
Description: CL/F was calculated as Dose/AUCinf.
Time Frame: Pre-dose,1, 2, 4, 6 and 8 hours post dose on C1D15
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 3 | 3 | 2 | 7 | 1 | 3 | 4 | 2 | 4 | 6
L/hr
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 4.07 and 4.72 L/hr. | 9.793 (0.82403) | 12.20 (1.2767) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 4.20 and 13.2 L/hr. | 13.14 (7.2301) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 67.9 L/hr. | 7.147 (2.8564) | 6.480 (2.3107) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 4.57 and 10.5 L/hr. | 8.138 (1.7244) | 11.18 (4.1290)
  Binimetinib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 2 | 4 | 6
  Binimetinib |  |  |  |  |  |  | 18.27 (6.4034) | 22.42 (20.947) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 9.75 and 23.9 L/hr. | 18.60 (2.5073) | 22.54 (10.178)

24. Secondary Outcome: Vz/F of PF-07284890 and Binimetinib for Multiple Dose: Phase 1a
Description: as for outcome 18
Time Frame: Pre-dose,1, 2, 4, 6 and 8 hours post dose on C1D15
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 1 | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2 | 2 | 1
Litre
  PF-07284890: number analyzed (Participants) | 1 | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2 | 2 | 0
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 50.6 L. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 59.5 and 141 L. | 126.4 (64.519) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 44.2 L. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 86.4 L. |  |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 49.8 L. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value were 28.1 and 53.9 L. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value were 35.7 and 50.1 L. |
  Binimetinib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Binimetinib |  |  |  |  |  |  |  |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 85.9 L. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 57.0 L. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 52.5 L.

25. Secondary Outcome: t½ of PF-07284890 and Binimetinib for Multiple Dose: Phase 1a
Description: T1/2 was calculated as loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. In the determination of the t1/2, steady-state was assumed and the pre-dose value was used for the 24-hour post-dose value, which could have enabled the reporting of the t1/2 value higher than 8 hours.
Time Frame: Pre-dose (24 hours post-dose concentration), 1, 2, 4, 6 and 8 hours post dose on C1D15
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 1 | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2 | 2 | 1
Hours
  PF-07284890: number analyzed (Participants) | 1 | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2 | 2 | 0
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 8.63 hours. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values were 4.54 and 9.15 hours. | 7.430 (4.1000) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 2.32 hours. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 4.17 hours. |  |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 3.80 hours. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value were 3.56 and 4.27 hours. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value were 3.37 and 4.23 hours. |
  Binimetinib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Binimetinib |  |  |  |  |  |  |  |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 2.49 hours. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 1.88 hours. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 3.98 hours.

26. Secondary Outcome: Accumulation Ratio (Rac) of PF-07284890 and Binimetinib for Multiple Dose: Phase 1a
Description: Rac was defined as area under the plasma concentration-time curve over the dosing interval at steady state (AUCss,τ) divided by area under the plasma concentration-time curve over the dosing interval from a single dose (AUCsd,τ).
Time Frame: Pre-dose,1, 2, 4, 6 and 8 hours post dose on C1D1 and C1D15
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 2 | 3 | 0 | 1 | 0 | 2 | 4 | 1 | 4 | 5
Ratio
  PF-07284890: number analyzed (Participants) | 2 | 2 | 3 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 2
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual (ratios) were 1.16 and 1.48. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual (ratios) were 0.435 and 1.02. | 1.024 (0.11484) |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual (ratio) was 2.22. |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual (ratios) were 0.583 and 2.21. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual (ratio) was 1.65. | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual (ratio) was 1.13. |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual (ratios) were 1.49 and 1.59.
  Binimetinib: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 4 | 5
  Binimetinib |  |  |  |  |  |  | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual (ratio) was 2.57. | 1.609 (0.54869) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual (ratio) was 2.87. | 1.950 (0.53560) | 2.088 (1.0472)

27. Secondary Outcome: Extracranial Response Rate by RECISTv1.1: Phase 1a
Description: Extracranial response rate was defined as the percentage of participants with a BOR of CR or confirmed PR in extracranial lesions by Investigator assessment per RECIST v1.1. CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (non-target) must have reduction in short axis to < 10 mm. PR: at least a 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of first dose until CR or PR (maximum treatment exposure: 542 days)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 6 | 2 | 4 | 4 | 1 | 3 | 5
Percentage of participants | 0 [0.0 to 84.2] | 0 [0.0 to 84.2] | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 45.9] | 0 [0.0 to 84.2] | 0 [0.0 to 60.2] | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8] | 0 [0.0 to 52.2]

28. Secondary Outcome: Intracranial Response Rate by mRECISTv1.1: Phase 1a
Description: Intracranial response rate as assessed using modified mRECIST v 1.1., was defined as the percentage of participants with brain or CNS involvement who achieved a CR or PR. CR: disappearance of all target and non-target lesions. For target lesions: Any pathological lymph nodes must be <10 mm in the short axis. For non-target lesions: All lymph nodes identified as a site of disease at baseline must be non-pathological (eg, <10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of first dose until CR or PR (maximum treatment exposure: 542 days)
Population: Intracranial response evaluable set included all participants enrolled and received at least one dose of study treatment and had measurable brain tumor at baseline and at least one post baseline intracranial assessment. Here "Overall Number of Participants Analyzed" as "0" signifies there was no participant evaluable in specified analysis set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 1 | 1 | 0 | 3 | 2 | 1 | 1 | 0 | 1 | 2 | 3
Percentage of participants | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] |  | 0 [0.0 to 70.8] | 0 [0.0 to 84.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] |  | 0 [0.0 to 97.5] | 0 [0.0 to 84.2] | 0 [0.0 to 70.8]

29. Secondary Outcome: ORR by RECISTv1.1: Phase 1a
Description: as for outcome 10
Time Frame: From date of first dose until CR or PR (maximum treatment exposure: 542 days)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 6 | 3 | 4 | 4 | 1 | 3 | 5
Percentage of participants | 0 [0.0 to 84.2] | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 45.9] | 0 [0.0 to 70.8] | 0 [0.0 to 60.2] | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8] | 0 [0.0 to 52.2]

30. Secondary Outcome: Overall Response Rate as Per RANO for Brain Tumours: Phase 1a
Description: RANO response rate was defined as the percentage of glioblastoma participants who achieved a CR or PR per RANO. CR was defined as complete disappearance of all enhancing measurable and non-measurable disease sustained for >= 4 weeks; no new lesions; stable or improved non-enhancing (T2/FLAIR) lesions; off steroids and neurological condition stable or improved. PR was defined as >=50% decrease compared to baseline in the sum of the perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks; no progression of non-measurable disease; stable or improved non enhancing (T2/FLAIR) lesions on the same or lower dose of corticosteroids compared with baseline scan; the corticosteroid dose at the time of the scan evaluation should be no greater than the dose at the time of the baseline scan and neurological condition stable or improved.
Time Frame: From date of first dose until CR or PR (maximum treatment exposure: 542 days)
Population: The response evaluable population included all participants who received at least one dose of study treatment and had measurable disease at baseline and at least one post baseline disease assessment. The outcome measure was to be evaluated only in glioblastoma participants. "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome and "0" represents no glioblastoma participants for respective reporting arms.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 2
Percentage of participants |  |  |  |  | 0 [0.0 to 70.8] |  |  |  | 100.0 [2.5 to 100.0] |  | 0 [0.0 to 84.2]

31. Secondary Outcome: Number of Participants With TEAEs, Serious TEAEs, Serious Treatment Related TEAEs, Grade 3 or 4 TEAEs and Grade 5 TEAEs by NCI CTCAE v5.0: Phase 1b
Description: An AE was any untoward medical occurrence in participant/ clinical study participant temporally associated with use of study intervention, whether/ not considered related to study intervention. TEAEs were defined as any AE that occurs during on-treatment period. The on-treatment period was defined as period that starts with first dose of study treatment and ends at last dose of study treatment +30 days, or start of new anti-cancer therapy [- 1 day], whichever occurred first. Serious TEAEs were any untoward medical occurrence at any dose that: suspected to cause death; life-threatening; required hospitalization; persistent/significant disability/incapacity and might caused congenital anomaly/birth defect. Serious treatment related TEAEs were related to study treatment and relatedness was judged by investigator. TEAEs were graded according to NCI-CTCAE v 5.0 (grade 3= severe, grade 4= life-threatening and grade 5= death related to AE). AEs included SAEs and all non-SAE.
Time Frame: From first dose of study treatment (Day 1) up to 30 days post last dose of study treatment/start of new anti-cancer therapy (-1 Day) whichever occurred first (maximum treatment exposure: 400 days, maximum follow up: 430 days)
Population: The safety analysis set included all enrolled participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 4 | 1 | 11
Participants
  Participants with TEAEs | 1 | 4 | 1 | 11
  Participants with Serious TEAEs | 0 | 3 | 0 | 3
  Participants with Serious Treatment-Related TEAEs | 0 | 1 | 0 | 0
  Participants with Grade 3 or 4 TEAEs | 0 | 3 | 0 | 6
  Participants with Grade 5 TEAEs | 0 | 1 | 0 | 1

32. Secondary Outcome: Number of Participants With Hematology Laboratory Abnormalities: Phase 1b
Description: The following hematology laboratory parameters were assessed: activated partial thromboplastin time prolonged, anemia, hemoglobin increased, INR increased, leukocytosis, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased and white blood cell decreased. Laboratory abnormality events were graded according to NCI CTCAE v5.0; grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening consequences and grade 5=death. In this outcome measure, those number of participants are reported who had hematology laboratory abnormality in any parameter of any CTCAE Grades.
Time Frame: From first dose of study treatment (Day 1) up to 30 days post last dose of study treatment (maximum treatment exposure: 400 days, maximum follow up: 430 days)
Population: The safety analysis set included all enrolled participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 4 | 1 | 11
Participants | 1 | 4 | 1 | 11

33. Secondary Outcome: Number of Participants With Chemistry Laboratory Abnormalities: Phase 1b
Description: The following chemistry laboratory parameters were assessed: alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, CPK increased, creatinine increased, hypercalcemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia and hyponatremia. Laboratory abnormality events were graded according to NCI CTCAE v5.0; grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening consequences and grade 5=death. In this outcome measure, those number of participants are reported who had chemistry laboratory abnormality in any parameter of any CTCAE Grades.
Time Frame: as for outcome 32
Population: The safety analysis set included all enrolled participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 4 | 1 | 11
Participants | 1 | 4 | 1 | 11

34. Secondary Outcome: Number of Participants With Dose Interruptions Due to TEAEs: Phase 1b
Description: as for outcome 5
Time Frame: During study treatment (from first dose of study treatment [Day 1] up to last dose of study treatment [maximum treatment exposure: 400 days])
Population: The safety analysis set included all enrolled participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 4 | 1 | 11
Participants | 0 | 4 | 0 | 8

35. Secondary Outcome: Number of Participants With Dose Reduction Due to TEAEs: Phase 1b
Description: as for outcome 6
Time Frame: as for outcome 34
Population: The safety analysis set included all enrolled participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 4 | 1 | 11
Participants | 0 | 1 | 0 | 2

36. Secondary Outcome: Number of Participants With Dose Discontinuations Due to TEAEs: Phase 1b
Description: In this outcome measure, dose discontinuations for any drug due to TEAEs were considered.
Time Frame: as for outcome 34
Population: The safety analysis set included all enrolled participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 4 | 1 | 11
Participants | 0 | 2 | 0 | 3

37. Secondary Outcome: Cmax of PF-07284890 and Binimetinib for Single Dose: Phase 1b
Time Frame: Pre-dose,1, 2, 4, 6, 8 and 24 hours post-dose on C1D1
Population: TThe PK parameter analysis population included all enrolled participants treated who did not have protocol deviations influencing PK parameter assessment, and have sufficient information to estimate at least 1 of the PK parameters of interest. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and contributed to data; 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 3 | 1 | 9
ng/mL
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 4730 ng/mL. | 3730 (639.06) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 7380 ng/mL. | 3406 (1558.8)
  Binimetinib: number analyzed (Participants) | 1 | 3 | 1 | 6
  Binimetinib | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 416 ng/mL. | 400.0 (120.65) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 748 ng/mL. | 387.2 (168.62)

38. Secondary Outcome: Tmax of PF-07284890 and Binimetinib for Single Dose: Phase 1b
Time Frame: Pre-dose,1, 2, 4, 6, 8 and 24 hours post-dose on C1D1
Population: as for outcome 13
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 3 | 1 | 9
Hours
  PF-07284890 | NA [NA to NA] — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence median and full range not reported. Individual value was 2.17 hours. | 2.25 [2.08 to 4.00] | NA [NA to NA] — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence median and full range not reported. Individual value was 4.07 hours. | 3.88 [2.00 to 4.08]
  Binimetinib: number analyzed (Participants) | 1 | 3 | 1 | 6
  Binimetinib | NA [NA to NA] — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence median and full range not reported. Individual value was 1.00 hours. | 1.25 [1.00 to 2.07] | NA [NA to NA] — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence median and full range not reported. Individual value was 2.18 hours. | 1.95 [0.917 to 3.82]

39. Secondary Outcome: AUClast of PF-07284890 and Binimetinib for Single Dose: Phase 1b
Description: AUClast was determined using the linear/log trapezoidal method.
Time Frame: Pre-dose,1, 2, 4, 6, 8 and 24 hours post-dose on C1D1
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 3 | 1 | 9
ng*hr/mL
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 19000 ng*hr/mL. | 9593 (1633.7) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 9890 ng*hr/mL. | 8033 (3703.1)
  Binimetinib: number analyzed (Participants) | 1 | 3 | 1 | 6
  Binimetinib | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 1360 ng*hr/mL. | 932.7 (208.62) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual value was 511 ng*hr/mL. | 967.7 (423.36)

40. Secondary Outcome: Cmax of PF-07284890 and Binimetinib for Multiple Dose: Phase 1b
Time Frame: Pre-dose,1, 2, 4, 6 and 8 hours post dose on C1D15
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 4 | 1 | 9
ng/mL
  PF-07284890: number analyzed (Participants) | 1 | 3 | 1 | 9
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 4730 ng/mL. | 2897 (925.00) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 7380 ng/mL. | 4301 (1647.6)
  Binimetinib: number analyzed (Participants) | 1 | 4 | 1 | 8
  Binimetinib | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 416 ng/mL | 557.5 (223.36) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 748 ng/mL. | 671.4 (380.67)

41. Secondary Outcome: Tmax of PF-07284890 and Binimetinib for Multiple Dose: Phase 1b
Time Frame: Pre-dose,1, 2, 4, 6 and 8 hours post dose on C1D15
Population: as for outcome 13
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 4 | 1 | 9
Hours
  PF-07284890: number analyzed (Participants) | 1 | 3 | 1 | 9
  PF-07284890 | NA [NA to NA] — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 3.87 hours. | 3.50 [1.75 to 3.92] | NA [NA to NA] — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 4.02 hours. | 2.08 [1.88 to 4.00]
  Binimetinib: number analyzed (Participants) | 1 | 4 | 1 | 8
  Binimetinib | NA [NA to NA] — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 0.983 hours. | 1.92 [1.00 to 3.97] | NA [NA to NA] — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 1.00 hours. | 1.50 [0.900 to 4.00]

42. Secondary Outcome: AUCtau of PF-07284890 and Binimetinib for Multiple Dose: Phase 1b
Time Frame: Pre-dose,1, 2, 4, 6 and 8 hours post dose on C1D15
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 4 | 1 | 9
ng*hr/mL
  PF-07284890: number analyzed (Participants) | 1 | 3 | 1 | 9
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 36300 ng*hr/mL. | 20130 (7072.0) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 65900 ng*hr/mL. | 31740 (13933)
  Binimetinib: number analyzed (Participants) | 1 | 4 | 1 | 8
  Binimetinib | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 2270 ng*hr/mL. | 2680 (408.00) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 3730 ng*hr/mL. | 3011 (1469.6)

43. Secondary Outcome: Cmin of PF-07284890 and Binimetinib for Multiple Dose: Phase 1b
Time Frame: Pre-dose,1, 2, 4, 6 and 8 hours post dose on C1D15
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 4 | 1 | 9
ng/mL
  PF-07284890: number analyzed (Participants) | 1 | 3 | 1 | 9
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 1310 ng/mL. | 755.7 (446.61) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 3490 ng/mL. | 1512 (947.80)
  Binimetinib: number analyzed (Participants) | 1 | 4 | 1 | 8
  Binimetinib | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 80.0 ng/mL. | 73.98 (31.319) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 146 ng/mL. | 120.4 (74.848)

44. Secondary Outcome: CL/F of PF-07284890 and Binimetinib for Multiple Dose: Phase 1b
Description: CL/F was calculated as Dose/AUCinf.
Time Frame: Pre-dose,1, 2, 4, 6 and 8 hours post dose on C1D15
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 4 | 1 | 9
L/hr
  PF-07284890: number analyzed (Participants) | 1 | 3 | 1 | 9
  PF-07284890 | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 8.26 L/hr. | 16.03 (4.7983) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 4.55 L/hr. | 11.02 (4.3338)
  Binimetinib: number analyzed (Participants) | 1 | 4 | 1 | 8
  Binimetinib | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 19.9 L/hr. | 17.13 (2.9273) | NA (NA) — As pre-specified in statistical analysis, statistics was to be provided only with >=3 evaluable measurements, hence mean and SD not reported. Individual values was 12.0 L/hr. | 21.19 (16.343)

45. Secondary Outcome: Intracranial Disease Control Rate (DCR) Per mRECIST v1.1: Phase1b
Description: DCR: percentage of participants with BOR of CR, PR/ SD, Non-CR/Non-PD by Investigator assessment. CR: disappearance of all target and non-target lesions. For target lesions: Any pathological lymph nodes must be <10 mm in short axis. For non-target lesions: All lymph nodes identified as site of disease at baseline must be non-pathological. PR: At least 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive disease (PD). PD: for target lesions- At least 20% increase in sum of diameters of target lesions, taking as reference smallest sum of diameters recorded since treatment started. In addition, sum must have an absolute increase of at least 5 mm. PD for non-target lesions- unequivocal progression of existing non-target lesions. Non-CR/Non-PD: persistence of 1/ more non-target lesion(s) identified as site of disease.
Time Frame: From date of first dose until CR or PR or SD (maximum treatment exposure: 400 days)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 2 | 1 | 3
Percentage of participants | 100.0 [2.5 to 100.0] | 50.0 [1.3 to 98.7] | 0 [0.0 to 97.5] | 100.0 [29.2 to 100.0]

46. Secondary Outcome: Overall Disease Control Rate (DCR) Per RECIST v1.1: Phase1b
Description: DCR: percentage of participants with BOR of CR, PR or SD, Non-CR/Non-PD by Investigator assessment. CR: disappearance of all target & non-target lesions. For target lesions: Any pathological lymph nodes must be <10 mm in short axis. For non-target lesions: All lymph nodes identified as site of disease at baseline must be non-pathological. PR: At least 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PD: for target lesions- At least 20% increase in sum of diameters of target lesions, taking as reference smallest sum of diameters recorded since treatment started. In addition, sum must have an absolute increase of at least 5 mm. PD for non-target lesions- unequivocal progression of existing non-target lesions. Non-CR/Non-PD: persistence of 1/ more non-target lesion(s) identified as site of disease.
Time Frame: From date of first dose until CR or PR or SD (maximum treatment exposure: 400 days)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 1 | 1 | 9
Percentage of participants | 100.0 [2.5 to 100.0] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 66.7 [29.9 to 92.5]

47. Secondary Outcome: Intracranial Progression Free Survival (PFS) by mRECISTv1.1: Phase1b
Description: PFS was defined as the time from date of the first dose of study treatment to the earliest documented disease progression by Investigator assessment, or death due to any cause, whichever occurred first. PD: for target lesions- At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters recorded since the treatment started . In addition, the sum must have an absolute increase of at least 5 mm. PD for non-target lesions- unequivocal progression of existing non-target lesions. If a participant had not had a PFS event at the time of the analysis cutoff or at the start of any new anticancer therapy, PFS was censored at the date of last adequate tumor assessment. Analysis was performed using Kaplan-Meier method.
Time Frame: From date of first dose of study treatment until first documentation of PD or death due to any cause or censoring date whichever occurred first (maximum treatment exposure: 400 days)
Population: The safety analysis set included all enrolled participants who received at least one dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 4 | 1 | 11
Months | NA [NA to NA] — Median and 95% Confidence Interval (CI) could not be calculated as participant did not have event. | NA [1.7 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated as there was only 1 participant evaluable with PFS of 1.4 months. | NA [4.1 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events.

48. Secondary Outcome: Overall Progression Free Survival (PFS): Phase1b
Description: PFS was defined as the time from date of the first dose of study treatment to the earliest documented disease progression by Investigator assessment, or death due to any cause, whichever occurred first. PD: for target lesions- at least 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (this includes baseline sum if that is smallest on study). In addition to the relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered a sign of progression. PD for non-target lesions- unequivocal progression of existing non-target lesion. If a participant had not had a PFS event at the time of the analysis cutoff or at the start of any new anticancer therapy, PFS was censored at the date of last adequate tumor assessment. Overall PFS included evaluation for brain metastasis and extracranial lesions. Analysis was performed using Kaplan-Meier method.
Time Frame: From start of study treatment until first documentation of PD or death due to any cause or censoring date (maximum treatment exposure: 400 days)
Population: The safety analysis set included all enrolled participants who received at least one dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 4 | 1 | 11
Months | NA [NA to NA] — Median and 95% CI could not be calculated as participant did not have event. | 1.7 [1.1 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated as there was only 1 participant evaluable with PFS of 1.4 months. | 4.1 [1.1 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events.

49. Secondary Outcome: Overall Survival (OS): Phase1b
Description: Overall survival was defined as the time from the date of first study treatment to the date of death due to any cause. Participants who were still alive at the end of the study or lost to follow-up were censored at the last date they were known to be alive. Analysis was performed using Kaplan-Meier method.
Time Frame: From start of study treatment until death due to any cause or censoring date (maximum treatment exposure: 400 days)
Population: The full analysis set includes all enrolled participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 4 | 1 | 11
Months | NA [NA to NA] — Median and 95% CI could not be calculated as participant did not had event. | 5.3 [1.1 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated as participant did not had event. | 12.1 [3.7 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events.

50. Secondary Outcome: Intracranial Duration of Response (DOR) by mRECIST v1.1: Phase1b
Description: DOR was defined as the time from date of the first radiographic response (CR or PR) to the earliest documented PD or death due to any cause. CR: disappearance of all target and non-target lesions. For target lesions: Any pathological lymph nodes must be <10 mm in the short axis. For non-target lesions: All lymph nodes identified as a site of disease at baseline must be non-pathological (eg, <10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD: for target lesions- At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters recorded since the treatment started. In addition, the sum must have an absolute increase of at least 5 mm. PD for non-target lesions- unequivocal progression of existing non target lesions.
Time Frame: From CR or PR until first documented PD or death due to any cause (maximum treatment exposure: 400 days)
Population: Intracranial response evaluable set included all participants enrolled and received at least one dose of study treatment and had measurable brain tumor at baseline and at least one post baseline intracranial assessment. Here "Overall Number of Participants Analyzed" as "0" signified participants did not have CR or PR.
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 0 | 0 | 0 | 0

51. Secondary Outcome: Overall DOR by RECIST v1.1: Phase1b
Description: DOR: time from date of first radiographic response (CR/PR) to earliest documented PD/ death due to any cause.CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (non-target) must have reduction in short axis to < 10 mm. PR: at least a 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD: for target lesions- At least 20% increase in sum of diameters of target lesions, taking as reference smallest sum of diameters recorded since treatment started. PD for non-target lesions- unequivocal progression of existing non-target lesions.
Time Frame: From CR or PR until first documented PD or death due to any cause (maximum treatment exposure: 400 days)
Population: The response evaluable population included all participants who received at least one dose of study treatment and had measurable disease at baseline and at least one post baseline disease assessment. Here "Overall Number of Participants Analyzed" signifies participants who have CR or PR and "0" signified participants did not have CR or PR for respective arms.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 0 | 0 | 1
Months | NA [NA to NA] — Since only 1 participant was evaluable hence median and 95% CI could not be calculated. Individual DOR was 11.3 months. |  |  | NA [NA to NA] — Since only 1 participant was evaluable hence median and 95%CI could not be calculated. Individual DOR was 8.38 months.

52. Secondary Outcome: Intracranial Time to Response (TTR) by mRECIST v1.1: Phase1b
Description: Time to response is the time from treatment start to date of first documentation of objective response (PR or CR). CR: disappearance of all target and non-target lesions. For target lesions: Any pathological lymph nodes must be <10 mm in the short axis. For non-target lesions: All lymph nodes identified as a site of disease at baseline must be non-pathological (eg, <10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of first dose until CR or PR (maximum treatment exposure: 400 days)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 2 | 1 | 3
Months | NA [NA to NA] — Median and 95%CI could not be estimated as participant (s) did not have event. | NA [NA to NA] — Median and 95%CI could not be estimated as participant (s) did not have event. | NA [NA to NA] — Median and 95%CI could not be estimated as participant (s) did not have event. | NA [NA to NA] — Median and 95%CI could not be estimated as participant (s) did not have event.

53. Secondary Outcome: Overall TTR by RECIST v1.1: Phase1b
Description: Time to response is the time from treatment start to date of first documentation of objective response (PR or CR). CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (non-target) must have reduction in short axis to < 10 mm. PR: at least a 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Response evaluable population.
Time Frame: From date of first dose until CR or PR (maximum treatment exposure: 400 days)
Population: The response evaluable population included all participants who received at least one dose of study treatment and had measurable disease at baseline and at least one post baseline disease assessment. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
Number analyzed (Participants) | 1 | 1 | 1 | 9
Months | NA [NA to NA] — Since only 1 participant was evaluable hence median and 95%CI could not be calculated. Individual TTR was 1.4 months. | NA [NA to NA] — Median and 95%CI could not be estimated as participant did not have an event. | NA [NA to NA] — Median and 95%CI could not be estimated as participant did not have an event. | NA [NA to NA] — Median and 95%CI could not be estimated as there were insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: From first dose of study treatment (Day 1) up to 30 days post last dose of study treatment/start of new anti-cancer therapy (-1 Day) whichever occurred first (For Phase 1a: maximum treatment exposure: 542 days; maximum follow-up: 572 days) and Phase 1b: (maximum treatment exposure: 400 days, maximum follow up: 430 days)
Description: Same event may appear as both non-SAE and SAE but are distinct events. An event may be categorised as serious in 1 subject and non-serious in another, or a subject may have experienced both SAE and non-SAE. The safety analysis set included all enrolled participants who received at least one dose of study intervention.
Groups:
- Phase 1a: PF-07284890 50 mg QD: Participants received PF- 07284890 50 milligrams (mg) oral dose once daily (QD) in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 100 mg QD: Participants received PF- 07284890 100 mg oral dose QD in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 200 mg QD: Participants received PF- 07284890 200 mg oral dose QD in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first
- Phase 1a: PF-07284890 200 mg BID: Participants received PF- 07284890 200 mg oral dose twice daily (BID) in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 300 mg BID: Participants received PF- 07284890 300 mg oral dose BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 450 mg BID: Participants received PF- 07284890 450 mg oral dose BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID: Participants received PF- 07284890 100 mg oral dose QD in combination with binimetinib 45 mg oral dose BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID: Participants received PF- 07284890 100 mg oral dose BID in combination with binimetinib 45 mg oral dose BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID: Participants received PF- 07284890 225 mg oral dose BID in combination with binimetinib 45 mg oral dose BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID: Participants received PF- 07284890 300 mg oral dose BID in combination with binimetinib 45 mg oral dose BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1b: Cohort 1: Cohort 1 included melanoma participants with asymptomatic brain metastases and no prior B-type Raf proto-oncogene (BRAF) inhibitor therapy. Participants received PF- 07284890 300 mg oral dose QD in combination with binimetinib 45 mg BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1b: Cohort 3: Cohort 3 included melanoma participants with asymptomatic brain metastases and with prior BRAF inhibitor therapy. Participants received PF- 07284890 300 mg oral dose QD in combination with binimetinib 45 mg BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1b: Cohort 4: Cohort 4 included melanoma participants with symptomatic brain metastases and with prior BRAF inhibitor therapy. Participants received PF- 07284890 300 mg oral dose QD in combination with binimetinib 45 mg BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
- Phase 1b: Cohort 5: Cohort 5 included participants with a mixture of tumor types, any brain disease and with or without prior BRAF inhibitor therapy. Participants received PF- 07284890 300 mg oral dose QD in combination with binimetinib 45 mg BID in a 21-day cycle. Participants continued treatment until disease progression, participant refusal, unacceptable toxicity, or up to 2 years, whichever occurred first.
Arm/Group | Phase 1a: PF-07284890 50 mg QD | Phase 1a: PF-07284890 100 mg QD | Phase 1a: PF-07284890 200 mg QD | Phase 1a: PF-07284890 200 mg BID | Phase 1a: PF-07284890 300 mg BID | Phase 1a: PF-07284890 450 mg BID | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID | Phase 1b: Cohort 1 | Phase 1b: Cohort 3 | Phase 1b: Cohort 4 | Phase 1b: Cohort 5
All-Cause Mortality (participants affected / at risk) | 1/2 | 4/4 | 0/3 | 2/3 | 4/10 | 2/3 | 2/4 | 3/4 | 1/2 | 4/5 | 4/8 | 0/1 | 3/4 | 0/1 | 4/11
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/4 | 0/3 | 3/3 | 4/10 | 2/3 | 1/4 | 1/4 | 1/2 | 2/5 | 3/8 | 0/1 | 3/4 | 0/1 | 3/11
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4 | 3/3 | 3/3 | 10/10 | 2/3 | 4/4 | 4/4 | 2/2 | 5/5 | 8/8 | 1/1 | 4/4 | 1/1 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a: PF-07284890 50 mg QD (N=2) | Phase 1a: PF-07284890 100 mg QD (N=4) | Phase 1a: PF-07284890 200 mg QD (N=3) | Phase 1a: PF-07284890 200 mg BID (N=3) | Phase 1a: PF-07284890 300 mg BID (N=10) | Phase 1a: PF-07284890 450 mg BID (N=3) | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID (N=4) | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID (N=4) | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID (N=2) | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID (N=5) | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID (N=8) | Phase 1b: Cohort 1 (N=1) | Phase 1b: Cohort 3 (N=4) | Phase 1b: Cohort 4 (N=1) | Phase 1b: Cohort 5 (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Jejunal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a: PF-07284890 50 mg QD (N=2) | Phase 1a: PF-07284890 100 mg QD (N=4) | Phase 1a: PF-07284890 200 mg QD (N=3) | Phase 1a: PF-07284890 200 mg BID (N=3) | Phase 1a: PF-07284890 300 mg BID (N=10) | Phase 1a: PF-07284890 450 mg BID (N=3) | Phase 1a: PF-07284890 100 mg QD + Binimetinib 45 mg BID (N=4) | Phase 1a: PF-07284890 100 mg BID + Binimetinib 45 mg BID (N=4) | Phase 1a: PF-07284890 150 mg BID + Binimetinib 45 mg BID (N=2) | Phase 1a: PF-07284890 225 mg BID + Binimetinib 45 mg BID (N=5) | Phase 1a: PF-07284890 300 mg BID + Binimetinib 45 mg BID (N=8) | Phase 1b: Cohort 1 (N=1) | Phase 1b: Cohort 3 (N=4) | Phase 1b: Cohort 4 (N=1) | Phase 1b: Cohort 5 (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 3
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Brugada syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Central serous chorioretinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dyschromatopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Serous retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subretinal fluid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 2 | 2 | 3 | 3 | 1 | 2 | 1 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 3 | 0 | 2 | 4 | 1 | 2 | 0 | 6
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 3 | 0 | 1 | 3 | 1 | 2 | 0 | 3
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 4 | 0 | 3 | 2 | 0 | 1 | 0 | 5
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ill-defined disorder (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 3
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1
Suprapubic pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 6
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Visual acuity tests (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 3 | 0 | 1 | 1 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Taste disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 4 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/88/NCT04543188/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT04543188/SAP_001.pdf